CLINICAL TRIAL: NCT07115654
Title: A Prospective Single-Arm Clinical Trial of BCMA/CD3 BsAb Therapy for POEMS Syndrome
Brief Title: BCMA/CD3 BsAb Therapy for POEMS Syndrome
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025047
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: POEMS Syndrome
Keywords: POEMS syndrome; Bispecific antibody
MeSH Terms: conditions — POEMS Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BsAbs-treatment group (Experimental)
  Interventions: Drug: CM336 (BCMA/CD3 bispecific antibody)

INTERVENTIONS:
Drug: CM336 (BCMA/CD3 bispecific antibody) — CM336 is a bispecific antibody targeting BCMA and CD3, designed to redirect T cells to eliminate abnormal plasma cells.

SUMMARY:
This is a prospective, single-arm, investigator-initiated clinical trial evaluating the safety and efficacy of a BCMA/CD3 bispecific antibody (CM336) in patients with POEMS syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosed with POEMS syndrome according to the 2025 Chinese Expert Consensus.
3. Deemed suitable for BCMA/CD3 bispecific antibody therapy by the investigator.
4. ECOG performance status 0-2.
5. Adequate organ function.
6. Provided written informed consent.

Exclusion Criteria:

1. Not meeting the diagnostic criteria for POEMS syndrome, including:

   * Chronic inflammatory demyelinating polyneuropathy (CIDP),
   * MGUS, multiple myeloma, amyloidosis, or other plasma cell disorders not meeting POEMS diagnostic criteria.
2. History of prior anti-plasma cell therapy, such as melphalan, cyclophosphamide, proteasome inhibitors, IMiDs, monoclonal antibodies, CAR-T, or bispecific antibodies (except:

   1. Immunosuppressants used for autoimmune neuropathy;
   2. Bisphosphonates used for bone disease;
   3. Topical or low-dose steroids ≤20 mg/day for rheumatic disease).
3. Investigator judges the patient unsuitable for BCMA/CD3 bispecific therapy (e.g., severe cardiopulmonary dysfunction).
4. Known allergy or intolerance to BCMA/CD3 bispecific antibody or any component.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Overall Response Rate (ORR) | Up to 12 months after treatment initiation
  To evaluate the safety and efficacy of BCMA/CD3 bispecific antibody therapy in patients with POEMS syndrome.

SECONDARY OUTCOMES:
Hematologic Response Rate | From treatment initiation to 3 months after end of treatment
VEGF Response Rate | From treatment initiation to 3 months after end of treatment
Duration of Response (DOR) | From first documented response to 6 months after end of treatment
Disease Control Rate (DCR) | From treatment initiation to 3 months after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided